CLINICAL TRIAL: NCT07075198
Title: Caesar Foot Take-Home Validation Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Hanger Clinic: Prosthetics & Orthotics (Other); WillowWood (Unknown); University of Hartford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13875; 1R44HD113432-01 (NIH)
Record Dates: First submitted 2025-06-24; First posted 2025-07-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Prosthesis User; Lower Limb Amputation Below Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Prosthesis Pre-Experimental Condition (Baseline) (No Intervention): The participant wears their usual prosthetic foot for 1 month before the experimental condition to collect baseline data.
- Caesar Foot (Experimental): The participant wears the Caesar Foot at home for about 2 months.
  Interventions: Device: Caesar Foot
- Usual Prosthesis Post-Experimental Condition (No Intervention): The participant wears their usual prosthetic foot for 1 month after completing the experimental condition and after receiving running training.

INTERVENTIONS:
Device: Caesar Foot — The investigators developed a bimodal, passive mechanical prosthetic foot called the Caesar Foot. The Caesar Foot has two modes: one optimized for walking, and one optimized for higher-energy activities like running. It has a switching device that was designed such that when it switches modes, it inherently accounts for the alignment and stiffness differences between walking and running feet (such as the longer length, higher stiffness, and different ground contact points required for running feet). Therefore, it should be largely comparable to a daily use prosthesis / walking foot when in walking mode, and an running specific prosthesis / running blade when in running mode. This foot is attached and aligned to the user's usual prosthetic socket.
  Arms: Caesar Foot

SUMMARY:
The rationale for this study is to conduct a take-home clinical trial to evaluate the impact of the bimodal Caesar foot in a real-world environment. Participants will take the device home and use it throughout their daily life for two months. A one-month baseline period, using their usual foot, will be completed both before and after the two-month period with the Caesar foot condition. Self-report surveys and performance-based measures will be collected in the clinic at the end of each condition. The intent of this study is to determine the Caesar foot's feasibility in a real-world environment. Data will be collected to understand impact to the user's daily life and physical activity through outcomes and participant feedback. The feedback obtained during this study will be essential to informing the design intended for commercialization.

DETAILED DESCRIPTION:
In this study, the investigators will administer a suite of performance-based and self-report measures to assess demonstrated and perceived differences between the foot conditions. The primary measure for this study is the Prosthetic Limb Users Survey of Mobility (PLUS-M). The investigators hypothesize that the participants will have greater mobility as reported by the PLUS-M in the Caesar foot as compared to their usual walking foot.

There are many aspects of mobility and activity that may not be captured by a single assessment. Therefore, the investigators will examine additional exploratory self-report measures after each condition during this pilot study, such as the PROMIS-Fatigue, PROMIS- Ability to Participate in Social Roles and Activities (PROMIS-APSRA), PLUS-Falls (PLUS-F), Trinity Amputation and Prosthesis Experience Scale - Revised (TAPES-R), EQ-5D, and custom surveys to further understand the participant's experiences and preferences with the Caesar foot. Surveys will be distributed on a HIPAA compliant platform, such as MS Forms, which can be completed on the clinic's laptop/tablet. Paper formats of the surveys may be distributed if issues arise with the online platform (e.g., internet outage).

The investigators will also conduct and collect performance-based measures from each participant, such as the 10-Meter Walk Test (10MWT), self-selected comfortable and fast gait speeds, comfortable running speed, and timed ¼ mile run. These measures are exploratory as well. The investigators will assess running effort objectively with the maximum heart rate (HRmax) during the ¼ mile run and subjectively using the Borg Rating of Perceived Exertion (RPE). During each 1-month take-home period, the investigators will measure participants' daily step count and track any falls that may occur.

In addition to wearing the activity monitor during the take-home periods, they will also be asked to participate in periodic calls with study team members to check in and report on any falls, issues they may be experiencing, and/or ask questions they may have about the study. These periodic calls will continue throughout the duration of the study.

As a pilot study, the goal of these measures is to better understand the impact of the Caesar foot on different aspects of a user's life and incorporate feedback into future designs.

The investigators plan to implement a pilot longitudinal comparative effectiveness study with an ABA study design, where A1 is the first control condition with the participant's usual prosthetic foot, B is the experimental condition with the Caesar Foot, and A2 is the second control condition with the participant's usual prosthetic foot. For each condition, the participant will use their usual prosthetic socket, and a certified prosthetist will set up and align them on the foot of interest. They will be provided time for acclimation to each prosthetic foot prior to Condition B and Condition A2 as they will have swapped to a foot that they were not using previously. Activity monitors will then be added to the prosthesis and the participant will wear the foot at home for one month.

All participants for this study will be individuals who desire to participate in running/jogging but do not currently have a running prosthesis, as determined by self-report. Eligible participants will be individuals who are at least 18 years of age and have transtibial limb absence of one or both limbs, a K-level of K3 or K4, the required foot size, weight, and limb clearance for one of the available Caesar prototypes, and have a well-fitting socket as determined by a certified prosthetist.

For the first month of the experimental condition (Condition B), the participant will wear the Caesar foot at home to acclimate to the foot and participate in a running training program. Training is necessary to fully utilize and maximize the performance with any prosthetic component. Therefore, the investigators leveraged the expertise of the investigators' collaborator, Alicia White, PT, DPT, ATC to implement a running training program. Dr. White developed the "Return to Run" program at the Department of Defense's Center for the Intrepid (CFI) to teach individuals with lower limb amputations how to run on a running blade prosthesis. She will train physical therapists at Hanger to teach study participants how to run on a prosthesis. Participants will attend at least two, but up to twelve, 1-hour training sessions.

The training will be designed to teach basic running mechanics that are agnostic of the foot used, as well as running blade-specific skills. The training will be tailored to the starting abilities of each participant and progress at an appropriate pace for each individual until they are competent at running (i.e., their running trainer deems they can safely run on the foot and the participant is comfortable doing so).

At a minimum, each participant will receive one training session to learn how to safely and properly run in the Caesar foot and a second session to demonstrate their competency in running with the foot. The participant will continue training until they show competence (as determined by their trainer) or until they receive twelve training sessions, whichever comes first. Because the participants will be new to running with a running foot, the training will be provided during the first month of condition B so participants can safely run on and acclimate to the Caesar Foot.

Participation in this study will consist of 5 site visits and about 4 months of at-home wear of the participant's usual foot and Caesar foot, as well as running training, and performance-based and self-report assessments throughout each condition. Participants may be asked to come in for additional visits for various reasons, such as technical issues with the device, running out of time in the visit before completing the outlined tasks/measures, etc.

Shortly after Visit 5, a study team member will conduct a final call with the participant to go over any other falls that may have occurred before Visit 5, clarify any missing data from surveys, and conduct the exit interview and preference survey. After this call, they will have completed their participation in study.

ELIGIBILITY:
Inclusion Criteria:

* Have transtibial limb absence of one or both limbs
* Express interest in running, but do not currently have a running blade (as determined by self-report)
* Are at least 18 years of age
* Are at least six months post amputation
* Are classified as K3 or K4 ambulator status as determined by a certified prosthetist
* Have an AMP score of at least 37
* Are capable of running safely as determined by a certified prosthetist's clinical judgement
* Have a well-fitting socket as determined by a certified prosthetist
* Have adequate clearance between distal end of the residual limb and ground for the Caesar foot
* Meets the foot size and weight class of one of the available Caesar prototypes

Exclusion Criteria:

* Present or sustained injuries to residual limb or contralateral leg affecting functional ability
* Non-English speaking participants will be excluded from this study due to limited access to interpreter services. These services would be needed for several visits, including training to learn how to use the device safely, along with requested verbal feedback from the participant to evaluate the design and usability of the system.
* Using a prosthetic foot that an individual is unfamiliar with for higher activity tasks may increase the risk of falling. Therefore, pregnant women should not participate in the study and will be screened by self-disclosure.

Individuals can be excluded at the discretion of the investigator for other unforeseen disqualifying criteria (such as specific cognitive issues, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Limb Users Survey of Mobility (PLUS-M) | 1 month
  The version of the PLUS-M being administered consists of 22 questions. Each question asks about their ability to ambulate in certain instances and at certain speeds, and is scored on a scale of 1 (unable to do) to 5 (without any difficulty). A higher score indicates a better outcome.
  This survey will be given at the end of each study condition. Since the first month of the Caesar condition will be for training and acclimation, the PLUS-M will be given after the second month that the participant is in the experimental condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johansson, Principal Investigator — Liberating Technologies, Inc.
Locations (1):
- Hanger Clinic, Austin, Texas, United States